CLINICAL TRIAL: NCT02605382
Title: Efficacy of 0.12% Chlorhexidine Gluconate for Non-surgical Treatment of Peri-implant Mucositis
Brief Title: Efficacy of 0.12% Chlorhexidine Gluconate for Peri-implant Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karyna de Melo Menezes, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRN
Record Dates: First submitted 2015-10-07; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Mucositis
Keywords: Dental Implantation; Chlorhexidine gluconate
MeSH Terms: conditions — Mucositis | interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- chlorhexidine gluconate (Experimental): 15 ml of solution every 12 hours, twice a day, 30 minutes after brushing, for 14 days
  Interventions: Drug: Chlorhexidine gluconate
- placebo (Placebo Comparator): 15 ml of solution every 12 hours, twice a day, 30 minutes after brushing, for 14 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Chlorhexidine gluconate
  Other Names: Chlorhexidine
  Arms: chlorhexidine gluconate
Drug: placebo — Solution chemical manufactured to mimic 0.12% chlorhexidine mouthwash
  Other Names: placebo solution
  Arms: placebo

SUMMARY:
The purpose of this study is to analyze the efficacy of 0.12% chlorhexidine gluconate as a chemical adjuvant for the treatment of peri-implant mucositis, in a non-surgical treatment protocol with a six-month follow-up.

DETAILED DESCRIPTION:
Determination of the sample size was based on the sample calculation for clinical trials, estimating a 50% success rate for the control group and 100% for the test group, which was then averaged for the two groups. With a standardized difference and power test of 85%, a total of 28 subjects per group were obtained.

Periapical radiographic examinations were performed before the collection of data to confirm the absence of bone loss, and threads exposition of the implants. The following clinical parameters were evaluated in both test and control groups; visible plaque index (VPI) and gingival bleeding index (GBI) were obtained for full mouth (IPV and ISG) and for each implant (VPI implant; GBI implant). For statistical purposes, percentages of faces with biofilm and marginal bleeding at teeth and implants were calculated. These parameters were evaluated at baseline and at one, three and six months post-therapy.

Keratinized mucosa width (KM), probing depth (PD implant), and bleeding on probing (BOP implant) were collected for all implants with a North Carolina periodontal probe at six sites. After data collection, an arithmetic averages of the sites with bleeding on probing, probing depths, and keratinized mucosa were calculated at baseline, three and six months. The peri-implant biotype for each implant was rated as thin or thick, according to probe transparency during probing depth.

Clinical parameters were collected by two operators, calibrated by the Kappa test for the keratinized mucosa, peri-implant biotype and probing depth.

After inclusion of the patients, anamnesis and initial examination were performed. The subjects were randomly divided, using a simple draw, in the following two groups: Test - (0.12% chlorhexidine digluconate associated with periodontal basic therapy) and Control - (placebo associated with periodontal basic therapy). Data were analyzed using descriptive and inferential statistics, with nonparametric tests, through a Statistical Package Social Sciences software (SPSS), version 17.0 (free version). The Friedman test was used for intragroup analysis and if any significant differences were observed, the Wilcoxon post-test was performed. Additionally, Mann-Whitney test was used for intergroup analysis. Chi-Square test was used to evaluate probing depth and bleeding on probing, according to the independent variables of interest: age, sex, treatment group, keratinized mucosa, peri-implant biotype, median VPI implant and GBI implant. Spearman correlation was also used to correlate probing depth and bleeding on probing after six months of follow-up. The implant was considered the unit of analysis and a value of p<0.05 was used to represent a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Systemically-healthy partially edentulous patients rehabilitated with functional dental implants and prostheses for at least 1 year;
* Patients had been diagnosed with peri-implant mucositis, probing depth up to 5 mm, bleeding on probing and no radiographic evidence of bone loss beyond the first two threads of the implant.

Exclusion Criteria:

* Non-smokers and not in maintenance therapy;
* Periodontal treatment during the last six months;
* Have not used antimicrobial (systemic or topical), anti-inflammatory or immunosuppressive drugs during the six months preceding the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | baseline
Bleeding on probing | three months
Bleeding on probing | six months

SECONDARY OUTCOMES:
Probing depth | baseline and at three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno CV Gurgel, Doctor, Study Director — Universidade Federal do Rio Grande do Norte